CLINICAL TRIAL: NCT02959073
Title: Evaluation of a New Self-assessed, Home-based Symptom Score in Cat Allergic Patients
Acronym: HypoScore-2
Status: Terminated | Type: Observational
Why Stopped: Company's strategic reasons
Sponsor: University of Zurich (Other)
Collaborators: Ottawa Allery Research Corporation (Unknown)
Responsible Party: Sponsor
Other Study IDs: ZU-HypoScore-002
Record Dates: First submitted 2016-11-03; First posted 2016-11-08 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Cat Allergy
Keywords: Symptom recording

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Symptom Recording — Subjects muss record their allergic symptoms after contact with their cats

SUMMARY:
In the last decades the prevalence of allergies has reached epidemic proportions. 10 to 15% of the population suffers from cat allergy. Investigators perform this study in order to further investigate symptom records and their evaluation in cat allergic patients.

Investigators primarily aim to better standardize the symptom recording of cat allergic persons under real-life conditions and to evaluate the effect of hypoallergenic cats on symptom strength.

ELIGIBILITY:
Inclusion Criteria:

* Participant understands the nature, meaning and scope of the study.
* Signed Informed Consent after being informed.
* Male and Female patients 18 years to 65 years of age.
* Positive screening prick test (mean wheal diameter equal or greater 3 mm) when tested with already standardized cat allergen extract.
* Positive screening prick test (wheal diameter equal or greater 3mm) to Histamine dihydrochloride 10 mg/ml.
* Positive Scratch Test when tested with cat dander sample of participant's cat.
* Baseline symptoms with a severity of "1" in at least 2 different symptoms.
* Owner of a cat that lives in the same household.
* Cat will not have been washed in the 4 weeks before starting the test phase.

Exclusion Criteria:

* Impaired in understanding the nature, meaning and scope of the study or incapable of giving written informed consent
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study
* Positive skin reaction in the prick test to negative control
* History of anaphylactic reaction to pet allergens
* Severe diseases influencing the results of the present study by discretion of the investigator
* Immunotherapy with fel d 1 / cat allergen preparation during the past two years
* Skin lesions and excessive hair-growth in the skin test areas
* Treatment with prohibited concomitant medications according to section 8.3 with the exception of medications with local effects which will not influence the results of the skin tests and the results of the other tests (testing period).
* The patient should not suffer from other respiratory allergies during this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy male or female participants with age between 18 and 65 years who suffer from confirmed cat allergy. The participants have to own a cat in the house/flat where they live.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Duration of provocation test under 2 different conditions | up to 9 weeks
Number of score Points resulting from symptom record | up to 9 weeks
fel d 1 concentration in cat dander | up to 9 weeks
  by collecting cat's fur
fel d 1 concentration in the air | up to 9 weeks
  by means of electrostatic dust collectors papers

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Senti Senti, Prof. Dr., Study Director — Hypo Pet AG, c/o University of Zurich
Locations (1):
- Ottawa Allergy Research Corporation (OARC), Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No